CLINICAL TRIAL: NCT06346249
Title: Workplace Based Physiotherapy of Elderly-care Workers With Non-specific Neck Pain: a Five Week Intervention With a One Month Follow-up Study.
Brief Title: Workplace Based Physiotherapy of Elderly-care Workers With Non-specific Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Mª Ángeles Cardero Durán, Principal Investigator, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49/2024
Record Dates: First submitted 2024-03-12; First posted 2024-04-04 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-02

CONDITIONS: Neck Pain
Keywords: non specific pain; physiotherapy; manual therapy; electrical stimulation therapy; therapeutic exercise
MeSH Terms: conditions — Neck Pain | interventions — Electric Stimulation Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The overall objective of this study is to determine the efficacy of a physical therapy intervention based on manual therapy, therapeutic exercise and application of electrical stimulation therapy in healthcare workers with non-specific neck pain.
  Interventions: Other: Electrical Stimulation Therapy; Other: Manual Therapy; Other: Exercise Therapeutic
- Control Group (No Intervention): The control group will not undergo any physiotherapy treatment therapy for neck pain.

INTERVENTIONS:
Other: Electrical Stimulation Therapy — Ten Electrical Stimulation Therapy sessions lasting 30 minutes were carried out. Analgesic currents of the TENS type, placed in the cervical region.
  Arms: Experimental Group
Other: Manual Therapy — Manual Therapy consistin of soft tissue mobilization and release techniques over the neck and craniocervical regions. Ten sessions.
  Arms: Experimental Group
Other: Exercise Therapeutic — The exercise therapeutic program consisting of neck movement control and stretching exercise. Ten sessions.
  Arms: Experimental Group

SUMMARY:
The overall objective of this study is to determine the efficacy of a physical therapy intervention based on manual therapy, therapeutic exercise and application of electrotherapy in healthcare workers with non-specific neck pain.

DETAILED DESCRIPTION:
The subjects included in the sample will be evaluated according to the aforementioned parameters by researchers trained and assigned for this purpose.

The data collection of the different variables will be performed before and after the completion of the program designed for the study. The physiotherapy intervention for the experimental group will have a duration of 10 sessions, twice a week.

ELIGIBILITY:
IInclusion Criteria:

* Age range between 18-60 years.
* Cervical pain of non-specific origin or Cervicalgia type I and II according to the Quebec - Task Force on Spinal Disorders.
* Be willing to participate in the study and sign the informed consent form.
* Have at least one year of seniority in the company exercising the current professional activity within the team of socio-health personnel.

Exclusion Criteria:

* Cervicalgia with neurological involvement or caused by pathologies such as: inflammatory disease, neurological disease, rheumatic disease, severe osteoporosis, fracture, dislocation, vertebro-basilar insufficiency, neoplasia or infection.
* Spine surgery.
* Present metallic implants at the spinal column level.
* Have received physiotherapy or alternative treatment in the last 6 months before starting the study.
* To present any type of inconvenience to the application of electrotherapy (score ≥45 points in EAPP).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in Pain | 5 weeks
  A visual analog scale (VAS). The scale is represented by a 10-centimeter line at the ends of which there are two adjectives whose ends there are two adjectives, absence of pain (0) and unbearable pain (10). The higher the score, the greater the pain.
Changes Pressure Pain | 5 weeks
  Pressure Pain with Algometry. To assess the mechanosensitivity of the trigger points , the pain threshold was measured at the pressure.
  Unit of measure Kg/cm2.
Changes in Disability | 5 weeks
  Neck Disability Index ( NDI) through which will give us the degree of disability neck pain.The NDI consists of 10 sections, 4 of them are related to subjective symptoms (pain intensity, headache, head, ability to concentrate and quality of sleep) and the other 6 are related to basic activities of daily living (ABVD) (personal care, ability to lift weights, reading, work, driving, leisure activities and free time). Each of the sections presents 6 possible answers, scoring these from 0 to 5 according to the progression of functional disability.

SECONDARY OUTCOMES:
Changes in Range of Motion | 5 weeks
  Measurement of joint amplitude with goniometry. The Range of Motion (ROM) exploration was performed with the subjects in sitting in order to stabilize the pelvis and the thoracic-lumbar spine. From this position, the degrees of maximum position reached by the subjects in each of the 6 movements of space.
  Unit of measurement in degrees of articulation.
General Health. | 5 weeks
  The Physical and Mental Health summary scales-12 (SF-12) contains 12 questions distributed in each of the 8 dimensions. The higher the score, the better the state of health.

CONTACTS AND LOCATIONS:
Overall Officials: María de los Ángeles Cardero Durán, Doctor, Principal Investigator — Universidad de Extremadura
Locations (1):
- María de los Ángeles Cardero Durán, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guzman J, Hurwitz EL, Carroll LJ, Haldeman S, Cote P, Carragee EJ, Peloso PM, van der Velde G, Holm LW, Hogg-Johnson S, Nordin M, Cassidy JD; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. A new conceptual model of neck pain: linking onset, course, and care: the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S14-23. doi: 10.1097/BRS.0b013e3181643efb. PMID 18204387
- [Background] de Campos TF, Maher CG, Steffens D, Fuller JT, Hancock MJ. Exercise programs may be effective in preventing a new episode of neck pain: a systematic review and meta-analysis. J Physiother. 2018 Jul;64(3):159-165. doi: 10.1016/j.jphys.2018.05.003. Epub 2018 Jun 19. PMID 29908853
- [Background] Nyman T, Grooten WJ, Wiktorin C, Liwing J, Norrman L. Sickness absence and concurrent low back and neck-shoulder pain: results from the MUSIC-Norrtalje study. Eur Spine J. 2007 May;16(5):631-8. doi: 10.1007/s00586-006-0152-6. Epub 2006 Jun 2. PMID 16741741
- [Background] Heintz MM, Hegedus EJ. Multimodal management of mechanical neck pain using a treatment based classification system. J Man Manip Ther. 2008;16(4):217-24. doi: 10.1179/106698108790818260. PMID 19771194
- [Background] Carroll LJ, Hogg-Johnson S, Cote P, van der Velde G, Holm LW, Carragee EJ, Hurwitz EL, Peloso PM, Cassidy JD, Guzman J, Nordin M, Haldeman S; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Course and prognostic factors for neck pain in workers: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S93-100. doi: 10.1097/BRS.0b013e31816445d4. PMID 18204406
- [Background] Driessen MT, Proper KI, van Tulder MW, Anema JR, Bongers PM, van der Beek AJ. The effectiveness of physical and organisational ergonomic interventions on low back pain and neck pain: a systematic review. Occup Environ Med. 2010 Apr;67(4):277-85. doi: 10.1136/oem.2009.047548. PMID 20360197
- [Background] Hidalgo B, Hall T, Bossert J, Dugeny A, Cagnie B, Pitance L. The efficacy of manual therapy and exercise for treating non-specific neck pain: A systematic review. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1149-1169. doi: 10.3233/BMR-169615. PMID 28826164
- [Background] Llamas-Ramos R, Pecos-Martin D, Gallego-Izquierdo T, Llamas-Ramos I, Plaza-Manzano G, Ortega-Santiago R, Cleland J, Fernandez-de-Las-Penas C. Comparison of the short-term outcomes between trigger point dry needling and trigger point manual therapy for the management of chronic mechanical neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Nov;44(11):852-61. doi: 10.2519/jospt.2014.5229. Epub 2014 Sep 30. PMID 25269764
- [Derived] Cardero Duran MLA, Espejo Antunez L, Fernandez Morales C, Albornoz Cabello M, Rodriguez Mansilla J. Workplace-Based Physiotherapy of Elderly Care Workers With Nonspecific Chronic Neck Pain: A Randomized Controlled Trial. J Occup Environ Med. 2026 Feb 1;68(2):e172-e181. doi: 10.1097/JOM.0000000000003566. Epub 2025 Oct 3. PMID 41042388

DOCUMENTS (1):
  • Informed Consent Form (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT06346249/ICF_000.pdf